CLINICAL TRIAL: NCT00058929
Title: A Multicenter, Randomized, Parallel Placebo-Controlled Study of the Safety and Efficacy of Subcutaneous Remodulin® Therapy After Transition From Flolan® in Patients With Pulmonary Arterial Hypertension
Brief Title: A Transition Study From Flolan® to Remodulin® in Patients With Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P01:13
Record Dates: First submitted 2003-04-14; First posted 2003-04-16 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Pulmonary Arterial Hypertension; Pulmonary Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: treprostinil sodium

SUMMARY:
This trial is a study of Remodulin in patients with pulmonary arterial hypertension who have been transitioned from Flolan therapy. The study consists of Screening, Baseline and Treatment Phases.

Patients meeting all inclusion/exclusion criteria during the Screening Phase will enter the Baseline Phase, during which baseline exercise capacity, vital signs, and clinical signs and symptoms of the disease will be assessed. After confirmation of all inclusion/exclusion criteria, patients will be assigned to study drug (Remodulin or placebo) and will enter the Treatment Phase. The Treatment Phase begins with a Dose Transition Period, during which patients will begin receiving subcutaneous study drug at a low dose determined by the patient's current dose of Flolan. The study drug dose will be increased gradually while the Flolan dose is decreased gradually over a period of up to 14 days. The dose changes will continue until Flolan therapy has been discontinued and the patient is stable on study drug.

Patients who are transitioned off Flolan, who are stable on study drug will be discharged from the clinic, and will continue to receive study drug on an outpatient basis. The patient will return to the clinic at Weeks 4 and 8 for assessments. Patients will remain on study drug for 8 weeks from the first dose of study drug. At Week 8, final assessments will be conducted and the patient will be dismissed from the study. Patients who successfully complete Week 8 assessments may be offered Remodulin therapy or other therapy, at the investigator's discretion.

DETAILED DESCRIPTION:
This trial is a multicenter, randomized, parallel placebo-controlled study of Remodulin in patients with pulmonary arterial hypertension with WHO Functional Class II or III clinical status who have been transitioned from Flolan therapy. The study consists of Screening, Baseline and Treatment Phases.

Patients meeting all inclusion/exclusion criteria during the Screening Phase will enter the Baseline Phase, during which baseline exercise capacity, vital signs, and clinical signs and symptoms of the disease will be assessed. After confirmation of all inclusion/exclusion criteria, patients will be randomized to study drug (1:1 Remodulin:placebo) and will enter the Treatment Phase. The Treatment Phase begins with a Dose Transition Period, during which patients will begin receiving subcutaneous study drug at a low dose determined by the patient's current dose of Flolan. The study drug dose will be increased gradually while the Flolan dose is decreased gradually over a period of up to 14 days. The dose changes will be done according to a recommended schedule, which may be modified if necessary according to the patient's clinical status. The dose changes will continue until Flolan therapy has been discontinued and the patient is stable on study drug, or until the patient has met the primary endpoint criteria.

Patients who are transitioned off Flolan, who are stable on study drug, and who have demonstrated the ability to properly self-administer study drug will be discharged from the clinic, and will continue to receive study drug on an outpatient basis. The patient will return to the clinic at Weeks 4 and 8 for assessments. At weeks other than Weeks 1, 4, and 8, the site staff will contact the patient to assess progress and adjust the study drug dose if necessary. Patients will remain on study drug for 8 weeks from the first dose of study drug. At Week 8, final assessments will be conducted and the patient will be dismissed from the study. Patients who successfully complete Week 8 assessments may be offered Remodulin therapy or other therapy, at the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria

Patients must:

* Be between 18 years and 75 years of age.
* If female, be physiologically incapable of childbearing or practicing an acceptable method of birth control.
* Have a current confirmed diagnosis of WHO Functional Class II or III pulmonary arterial hypertension (either PPH or PAH associated with the scleroderma spectrum of diseases).
* Have been clinically stable with regard to signs and symptoms of PAH for at least the last 30 days.
* Have a baseline six-minute walk distance of at least 250 meters.
* Have been receiving Flolan therapy for at least 6 months, and have documented clinical benefit from Flolan therapy on an exercise assessment.
* Be receiving Flolan at a dose of at least 15 ng/kg/min, but not more than 75 ng/kg/min, and have maintained the current dose of Flolan unchanged for at least 30 days at screening.
* Unless contraindicated, be able to receive one of the following anticoagulants: warfarin to achieve an INR between 2.0 and 3.0 or heparin to produce an aPTT between 1.3 to 1.5 times control, unless higher levels are clinically indicated.
* Be mentally and physically capable of learning to administer study drug using an subcutaneous infusion pump.

Exclusion Criteria

Patients must not:

* Be a nursing or pregnant woman (women of childbearing potential must have a negative serum pregnancy test).
* Have had a new type of chronic therapy (including but not limited to oxygen, a different category of vasodilator, a diuretic, digoxin) for pulmonary hypertension added within the last month.
* Have any pulmonary hypertension medication except for anticoagulants discontinued within the week prior to study entry.
* Have ever received Remodulin or any other prostaglandin/prostacyclin analog other than Flolan or Beraprost; or have received Bosentan or any other endothelin receptor antagonist within the past 30 days.
* Have evidence of significant parenchymal lung disease as evidenced by pulmonary function tests within the last six months as follows (any one of the following):

  1. Total Lung Capacity < 60% (predicted), or
  2. If Total Lung Capacity is between 60% and 70% (predicted), a High Resolution CT scan must be performed to document diffuse interstitial fibrosis or alveolitis, or
  3. FEV/FVC ratio < 50%, or

     * All Scleroderma patients must have Pulmonary Function Test performed within six weeks prior to study entry.
* Be positive for HIV.
* Have Portal Hypertension.
* Have a history of uncontrolled Sleep Apnea within the past three months.
* Have a history of left-sided heart disease including:

  1. Aortic or mitral valve disease or,
  2. Pericardial constriction or,
  3. Restrictive or congestive cardiomyopathy.
* Have evidence of current left-sided heart disease as defined by:

  1. PCWPm or left ventricular end diastolic pressure > 15 mmHg or
  2. LVEF < 40% by MUGA or Angiography or echocardiography or
  3. LV Shortening Fraction < 22% by echocardiography or
  4. Symptomatic coronary disease (demonstrable ischemia).
* Have any other disease that is associated with pulmonary hypertension (e.g. congenital systemic to pulmonary shunt, sickle cell anemia, schistosomiasis).
* Have a musculoskeletal disorder (e.g. arthritis, artificial leg, etc.) or any other disease, which is thought to limit ambulation, or be connected to a machine, which is not portable.
* Have uncontrolled systemic hypertension as evidenced by systolic blood pressure greater than 160 mmHg or diastolic blood pressure greater than 100 mmHg.
* Have used prescription appetite suppressants within 3 months of study entry.
* Have chronic renal insufficiency as defined by creatinine greater than 3.5 mg/dL or the requirement for dialysis.
* Be receiving an investigational drug, have in place an investigational device, or have participated in an investigational drug study within the past 30 days.
* Have had an atrial septostomy.
* Have anemia (hemoglobin <10 g/dL), active infection or any other ongoing condition that would interfere with the interpretation of study assessments.
* Have any serious or life-threatening disease other than conditions associated with PAH (e.g. malignancy requiring aggressive chemotherapy, renal dialysis, etc.).
* Have unstable psychiatric status or be mentally incapable of understanding the objectives, nature or consequences of the trial, or any condition which in the investigator's opinion would constitute an unacceptable risk to the patient's safety.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39
Dates: Start 2002-10; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of Southern California, Los Angeles, California
  - Harbor-UCLA Medical Center, Torrance, California
  - The Rush Heart Institute Center for Pulmonary Heart Disease, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Baylor College of Medicine, Houston, Texas
  - LDS Hospital, Salt Lake City, Utah